CLINICAL TRIAL: NCT05062343
Title: Cook Balloon vs Dilapan-S for Outpatient Cervical Ripening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Sarah E Little, Clinical Instructor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021P002625
Record Dates: First submitted 2021-09-09; First posted 2021-09-30 (Actual); Results first posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Induced; Birth
Keywords: Induction of labor; Cervical ripening

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Care Provider
Masking Description: Physician performing the cervical exams will be blinded to the patient's study arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Dilapan-S (Active Comparator): After randomization, the patient will have Dilapan-S placed via sterile speculum exam with placement of 3-5 rods. The rods will remain in place until expelled or up to 24 hours or until the scheduled return to labor and delivery. At presentation to labor and delivery, the rods will be confirmed expelled or will be removed and a blinded examiner will complete a sterile cervical exam. At that point the primary health care providers will manage further labor per their standard practice.
  Interventions: Device: Dilapan-S
- Cook Catheter (Active Comparator): After randomization, the patient will have the Cook catheter placed via sterile vaginal or speculum exam with the uterine component of the balloon inflated to maximum 60mL. The balloon will remain in place until expelled or up to 24 hours or until the scheduled return to labor and delivery. At presentation to labor and delivery, the Cook catheter will be confirmed expelled or will be removed and a blinded examiner will complete a sterile cervical exam. At that point the primary health care providers will manage further labor per their standard practice.
  Interventions: Device: Cook Cervical Ripening Balloon

INTERVENTIONS:
Device: Dilapan-S — Osmotic dilator
  Arms: Dilapan-S
Device: Cook Cervical Ripening Balloon — Double balloon catheter for cervical ripening
  Other Names: Cook catheter
  Arms: Cook Catheter

SUMMARY:
The goal of this study is to compare Cook balloon and Dilapan-S for outpatient cervical ripening to see if Dilapan-S is non-inferior in increasing Bishop score compared to the Cook balloon.

DETAILED DESCRIPTION:
Upon presentation for cervical ripening appointment, a sterile vaginal exam will be completed to assign Bishop score, as per standard routine. Once the patient has been consented and randomized, the participant will have a Cook catheter or Dilapan-S inserted. For the Cook catheter, the uterine component of the balloon will be inflated to maximum 60mL, the vaginal balloon will not be inflated per standard practice and per the literature that shows slightly increased pain and negligible improvement in cervical ripening. The catheter will be taped to the inner thigh with gentle traction. For Dilapan-S, 3-5 dilators will be placed.

After placement, the patient will be discharged home with strict return precautions per the outpatient cervical ripening protocol. Patients must return to labor and delivery within 24 hours of cervical ripening agent placement at their scheduled inpatient induction time.

Upon return to labor and delivery, if not already expelled, the mechanical ripening device will be removed, and an examiner blinded to the cervical ripening method will complete a sterile vaginal exam to assign a Bishop score.

At that point health care providers will manage active labor per usual practice. Labor interventions are at the discretion of the healthcare provider. The need for operative delivery or cesarean section will be at the discretion of the healthcare provider.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years of age
* Term (37-41 6/7 weeks gestational age)
* Low risk (i.e. without any maternal or fetal co-morbidity) and who are candidates for outpatient cervical ripening per the Brigham and Women's outpatient cervical ripening protocol
* Singleton pregnancy
* Cephalic presentation

Exclusion Criteria:

* Prior cesarean section
* Any contraindication to outpatient cervical ripening per Brigham and Women's outpatient cervical ripening protocol
* Non-English-speaking

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — All pregnancy patients
Enrollment: 80 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2023-07-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's HospitaL, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grobman WA, Rice MM, Reddy UM, Tita ATN, Silver RM, Mallett G, Hill K, Thom EA, El-Sayed YY, Perez-Delboy A, Rouse DJ, Saade GR, Boggess KA, Chauhan SP, Iams JD, Chien EK, Casey BM, Gibbs RS, Srinivas SK, Swamy GK, Simhan HN, Macones GA; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Labor Induction versus Expectant Management in Low-Risk Nulliparous Women. N Engl J Med. 2018 Aug 9;379(6):513-523. doi: 10.1056/NEJMoa1800566. PMID 30089070
- [Background] Saad AF, Villarreal J, Eid J, Spencer N, Ellis V, Hankins GD, Saade GR. A randomized controlled trial of Dilapan-S vs Foley balloon for preinduction cervical ripening (DILAFOL trial). Am J Obstet Gynecol. 2019 Mar;220(3):275.e1-275.e9. doi: 10.1016/j.ajog.2019.01.008. Epub 2019 Feb 18. PMID 30790569
- [Background] Ausbeck EB, Jauk VC, Xue Y, Files P, Kuper SG, Subramaniam A, Casey BM, Szychowski JM, Harper LM, Tita AT. Outpatient Foley Catheter for Induction of Labor in Nulliparous Women: A Randomized Controlled Trial. Obstet Gynecol. 2020 Sep;136(3):597-606. doi: 10.1097/AOG.0000000000004041. PMID 32769658
- [Background] Saunders SJ, Saunders R, Wong T, Saad AF. Out-of-Hospital Cervical Ripening With a Synthetic Hygroscopic Cervical Dilator May Reduce Hospital Costs and Cesarean Sections in the United States-A Cost-Consequence Analysis. Front Public Health. 2021 Jun 18;9:689115. doi: 10.3389/fpubh.2021.689115. eCollection 2021. PMID 34222185

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dilapan-S | Cook Catheter
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dilapan-S | Cook Catheter | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.8 (4.8) | 33.3 (4.1) | 32.5 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 80
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 11
  Not Hispanic or Latino | 34 | 34 | 68
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 2 | 8
  White | 27 | 33 | 60
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 3 | 7
Gestational age [Mean (Standard Deviation); unit: Weeks] | 39.4 (1.0) | 39.3 (0.7) | 39.4 (0.9)
Parity: Nulliparity, Multiparity [Count of Participants; unit: Participants] — Number of participants without a prior delivery (nulliparity) and with 1 more deliveries (multiparity)
  Participants
    Nulliparity | 28 | 28 | 56
    Multiparity | 12 | 12 | 24
Insurance type: public, private [Count of Participants; unit: Participants]
  Public insurance | 9 | 4 | 13
  Private insurance | 31 | 36 | 67

OUTCOME MEASURES:

1. Primary Outcome: Change in Bishop Score
Description: Difference in Bishop score calculated from exam at time of device removal minus Bishop score calculated from exam at time of device placement. Bishop score, or cervical score, ranges from a minimum of 0 to maximum of 13. Higher scores indicate that the cervix is more favorable, or ready for labor. Thus, change in Bishop score could range from -13 to +13 with a higher number showing more change in the score, or more cervical ripening.
Time Frame: Up to 24 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Dilapan-S | Cook Catheter
Number analyzed (Participants) | 40 | 40
score on a scale | 3.0 [2.0 to 5.0] | 3.0 [2.0 to 4.5]
Statistical Analysis 1: Comparison: Dilapan-S vs Cook Catheter; Test type: Superiority; p = 0.91, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Patient Satisfaction
Description: Patient Satisfaction score based on patient survey. Range from 0 (unsatisfied) to 10 (highly satisfied).
Time Frame: Assessed upon device removal, within 24 hours
Population: 3 participants did not fill out the survey and were not included in this outcome measure analysis.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Dilapan-S | Cook Catheter
Number analyzed (Participants) | 38 | 39
score on a scale | 9 [8 to 10] | 8 [5 to 9]
Statistical Analysis 1: Comparison: Dilapan-S vs Cook Catheter; Test type: Superiority; p < 0.01, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Mode of Delivery: Vaginal Delivery, Cesarean Delivery
Description: Mode of delivery, vaginal (including spontaneous vaginal, forceps and vacuum) and cesarean delivery
Time Frame: Assessed at the time of delivery, within 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Dilapan-S | Cook Catheter
Number analyzed (Participants) | 40 | 40
Participants
  Vaginal delivery | 30 | 30
  Cesarean delivery | 10 | 10
Statistical Analysis 1: Comparison: Dilapan-S vs Cook Catheter; Test type: Superiority; p = 1.0, Chi-squared

4. Secondary Outcome: Time on Labor and Delivery
Description: Time from admission on labor and delivery until delivery. Measured in hours.
Time Frame: Assessed at the time of delivery, within 1 week
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Dilapan-S | Cook Catheter
Number analyzed (Participants) | 40 | 40
Hours | 20.1 [13.9 to 26.2] | 17.0 [11.7 to 28.4]
Statistical Analysis 1: Comparison: Dilapan-S vs Cook Catheter; Test type: Superiority; p = 0.89, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Maternal Length of Stay
Description: Admission Date/Time to Discharge Date/Time
Time Frame: Assessed at end of study period (week 4)
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Dilapan-S | Cook Catheter
Number analyzed (Participants) | 40 | 40
Days | 3.2 [2.7 to 4.7] | 2.9 [2.7 to 3.9]
Statistical Analysis 1: Comparison: Dilapan-S vs Cook Catheter; Test type: Superiority; p = 0.98, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Cervical Ripening Success Score: No Failure, Failure
Description: Failure defined by: inability to place intervention agent or need for further cervical ripening after removal
Time Frame: Assessed at the time of device removal, within 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Dilapan-S | Cook Catheter
Number analyzed (Participants) | 40 | 40
Participants
  No failure | 33 | 25
  Failure | 7 | 15
Statistical Analysis 1: Comparison: Dilapan-S vs Cook Catheter; Test type: Superiority; p = 0.045, Chi-squared

7. Secondary Outcome: Composite Maternal Morbidity: Morbidity, no Morbidity
Description: Morbidity defined as any one of the following: higher-order laceration, blood transfusion, endometritis, wound infection, venous thromboembolism, hysterectomy, ICU admission or death
Time Frame: Assessed at end of study period (week 4)
Measure: Count of Participants; unit: Participants
Arm/Group | Dilapan-S | Cook Catheter
Number analyzed (Participants) | 40 | 40
Participants
  Morbidity | 8 | 8
  No Morbidity | 32 | 32
Statistical Analysis 1: Comparison: Dilapan-S vs Cook Catheter; Test type: Superiority; p = 1, Chi-squared

8. Secondary Outcome: Composite Neonatal Morbidity: Morbidity, no Morbidity
Description: Morbidity defined as any one of the following: culture-proven neonatal sepsis, neonatal blood transfusion, hypoxic-ischemic encephalopathy, intraventricular hemorrhage grade 3 or 4, or therapeutic hypothermia
Time Frame: Assessed at end of study period (week 4)
Measure: Count of Participants; unit: Participants
Arm/Group | Dilapan-S | Cook Catheter
Number analyzed (Participants) | 40 | 40
Participants
  Morbidity | 1 | 0
  No morbidity | 39 | 40
Statistical Analysis 1: Comparison: Dilapan-S vs Cook Catheter; Test type: Superiority; p = 1, Fisher Exact

ADVERSE EVENTS:
Time Frame: Events collected up until 6 weeks after delivery
Arm/Group | Dilapan-S | Cook Catheter
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-24): https://cdn.clinicaltrials.gov/large-docs/43/NCT05062343/Prot_SAP_000.pdf